CLINICAL TRIAL: NCT00005343
Title: Social Support and CHD Risk Factors--A Community Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4206
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To examine the mechanism through which social support affects morbidity and mortality from coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Two hypotheses have been proposed to account for the effects of social support on cardiovascular morbidity and mortality. Both hypotheses operate through effects on risk factors for coronary heart disease, specifically arterial blood pressure and serum lipids. The stress- buffering hypothesis states that social support functions as a social resource for individuals exposed to social stressors; those persons with more support are less vulnerable to the risk-enhancing effects of stressors. The health behavior hypothesis states that persons with more support engage in more positive health behaviors, such as avoiding tobacco; moderate alcohol use; exercise; and, a prudent diet. A major limitation in research to evaluate these alternative hypotheses has been the failure to conceptualize and measure social support in a way appropriate to detect its effects in varying social and cultural contexts. This is a major issue in research in sub-cultural communities that are also high risk communities, such as African-Americans.

DESIGN NARRATIVE:

A cross-sectional survey of social stressors, social supports, health behaviors, and arterial blood pressure and serum lipids was conducted in a Black community in the rural South to evaluate the relative strengths of the stress-buffering versus the health behavior hypothesis. Social support was measured using a culturally appropriate technique which was sensitive both to the distinction between kin and nonkin social support, and the modification of the effects of that support by generational status. Multiple regression analysis and path analysis were used to evaluate the alternative hypotheses.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01; Study Completion 1995-12

REFERENCES:
- [Background] Dressler WW. Social identity and arterial blood pressure in the African-American community. Ethn Dis. 1996 Winter-Spring;6(1-2):176-89. PMID 8882846
- [Background] Dressler WW. Hypertension in the African American community: social, cultural, and psychological factors. Semin Nephrol. 1996 Mar;16(2):71-82. PMID 8668863
- [Background] Dressler WW. Social status and the health of families: a model. Soc Sci Med. 1994 Dec;39(12):1605-13. doi: 10.1016/0277-9536(94)90074-4. PMID 7846557